CLINICAL TRIAL: NCT05942287
Title: The Effects of Obesity and Weight Loss in Heart Failure: Imaging the Obesity Paradox Using Magnetic Resonance Imaging and Spectroscopy - Heart Failure With Reduced Ejection Fraction Substudy
Brief Title: The Effect of Obesity and Weight Loss in Heart Failure With Reduced Ejection Fraction.
Acronym: SLEnDR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 161729 (D); 15/SC/0004 (Other: Research Ethics Committee)
Record Dates: First submitted 2023-07-03; First posted 2023-07-12 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure; Heart Failure With Reduced Ejection Fraction; Obesity; Overweight
Keywords: heart failure; weight loss; low energy diet; reduced ejection fraction
MeSH Terms: conditions — Heart Failure; Obesity; Overweight; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet intervention (Experimental): Diet intervention (in addition to standard clinical care)
  Interventions: Other: Diet intervention
- Standard clinical care (No Intervention): Standard clinical care only

INTERVENTIONS:
Other: Diet intervention — The diet intervention delivers a weight loss program. The main component is a total diet replacement low energy diet. The intervention includes a gradual food reintroduction phase and maintenance strategies.
  Arms: Diet intervention

SUMMARY:
This study looks at the effects of weight loss in people who have heart failure with reduced ejection fraction (HFpEF) and are overweight or obese.

The main questions it aims to answer are whether weight loss in this group of people improves:

* The heart's shape and how well it pumps blood
* The person's quality of life and how much they can exercise

Participants will attend 2 study visits, separated by 3-6 months. The intervention period takes place in between the 2 study visits.

Each study visit may involve measurements including:

Symptom and quality of life questionnaires Body measurements such as height and weight Blood tests Ultrasound scans of the heart (echocardiogram) Magnetic Resonance Imaging (MRI) scans of the heart 6 minute walk test Participants are randomly allocated (in other words, by lottery) to either 'diet' or 'control' groups. The control group will continue standard care.

The diet group will be enrolled in a weight loss program supervised by the study team. Participants in the diet group will replace their usual meals with meal replacement products specifically designed to deliver a low calorie diet for weight loss. The products will consist of formula soups, shakes and porridges. This diet would last 8 weeks, followed by a guided period of food reintroduction and maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure determined by left ventricular ejection fraction 20-45%
* Body mass index > 27.5kg/m^2

Exclusion Criteria:

* Contraindications to magnetic resonance imaging
* NYHA class IV
* Pregnancy, planned pregnancy or lactating
* Significant valvular, ischemic, infiltrative or other potentially confounding cardiac disease
* Any other conditions which may potentially compromise the safety or scientific validity of the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Left ventricular ejection fraction | Change from baseline at 3-6 months
  On cardiac magnetic resonance imaging (CMR)

SECONDARY OUTCOMES:
Body weight | Change from baseline at 3-6 months
Six minute walk distance | Change from baseline at 3-6 months
Kansas City Cardiomyopathy Questionnaire (KCCQ) | Change from baseline at 3-6 months
  A scale of 0 - 100, where higher scores indicate better outcomes.
N-terminal pro brain natriuretic peptide (NTproBNP) | Change from baseline at 3-6 months

OTHER OUTCOMES:
Left ventricular mass | Change from baseline at 3-6 months
  on CMR
Left atrial volume | Change from baseline at 3-6 months
  on CMR

CONTACTS AND LOCATIONS:
Overall Officials: Oliver J Rider, DPhil, Principal Investigator — University of Oxford
Locations (2):
- Jersey General Hospital, Jersey, Jersey, Jersey
- Jenny Rayner, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided